CLINICAL TRIAL: NCT04007666
Title: Leveraging Implementation Science to Increase Access to Trauma Treatment for Incarcerated Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 229172; K23DA048162 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-07-05 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Substance Use Disorders; Drug Abuse; Alcohol Abuse; Posttraumatic Stress Disorder; PTSD; Recidivism; Depression
Keywords: Incarcerated; Prisoners; Implementation Science
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Stress Disorders, Post-Traumatic; Recidivism; Depression | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Processing Therapy (CPT) (Experimental): CPT is a gold-standard evidence-based psychotherapy for PTSD that combines education about trauma with strategies to challenge the trauma-related cognitions that are theorized to maintain PTSD symptoms. It can be delivered in group and individual formats, but will be delivered in a group format in this project due to feasibility in the setting. Structure will be based on feedback obtained during completion of Aim 2 while remaining within the range evaluated in prior research (i.e., 8-12 sessions, 1-2x per week, each lasting 1.5-2 hours).
  Interventions: Behavioral: Cognitive Processing Therapy
- Coping Skills Group (Active Comparator): The Coping Skills Group will match for attention and dose, without adding any cost to the system. Exact content will be determined during completion of Aim 2; however, project sites already provide coping-focused programming and coping-skill approaches to trauma treatment are a common alternative to evidence-based therapies for PTSD, such as CPT, that deal more directly with the index trauma. To provide an enhanced standard of care, the investigator will review treatment materials (workbooks, handouts) already used in prison settings and arrange a curriculum of skills similar to those in coping-focused trauma-informed interventions (e.g., psychoeducation, assertiveness).
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy is an evidence-based psychotherapy for PTSD that combines education about trauma with strategies to challenge the trauma-related cognitions that are theorized to maintain PTSD symptoms.
  Other Names: CPT
  Arms: Cognitive Processing Therapy (CPT)
Behavioral: Control Group — Coping-focused treatment.
  Arms: Coping Skills Group

SUMMARY:
The unmet need for effective addiction treatment within the criminal justice system "represents a significant opportunity to intervene with a high-risk population" according to NIDA's 2016-2020 strategic plan. The plan also encourages the development and evaluation of implementation strategies that address the needs of the criminal justice system. The proposed research will be conducted as part of Dr. Zielinski's Mentored Patient-Oriented Research Career Development Award (K23), which aims to: 1) advance knowledge on implementation of a gold-standard psychotherapy for trauma, Cognitive Processing Therapy (CPT), in the prison setting and 2) examine whether prison-delivered CPT reduces drug use, psychiatric symptoms, and recidivism compared to a control condition (a coping-focused therapy). These foci have been selected because severe trauma exposure, substance use, and justice-involvement overwhelmingly co-occur in prison populations. The three specific aims in this research are: 1) Use formative evaluation to identify factors that may influence implementation and uptake of CPT in prisons, 2) Adapt CPT for incarcerated drug users and develop a facilitation-based implementation guide to support its uptake, and 3) conduct a participant-randomized Hybrid II trial to assess effectiveness and implementation outcomes of CPT with incarcerated drug users. Participants will include people who have been incarcerated (pre- and post-release from incarceration) and prison stakeholders who will be purposively sampled based on their role in implementation of CPT and other programs. Anticipated enrollment across all three Aims is 244 adult men and women.

ELIGIBILITY:
Inclusion criteria for all participants:

* 18 years of age or older
* Able to understand and speak English
* Able to give informed consent

Inclusion criteria for key stakeholders/informants participating in Aims 1-3 (additional requirements):

* All items listed in "Inclusion criteria for all participants"
* Invited by the PI to participate, due to specific role within project sites (e.g., current Warden, treatment staff member, officer, study therapist)

Inclusion criteria for prisoners completing formative evaluation interviews in Aim 1 and pre-treatment assessments in Aim 3 (additional requirements):

* All items listed in "Inclusion criteria for all participants"
* Incarcerated in either East Central Arkansas Community Correction Center (ECACCC) or Northeast Arkansas Community Correction Center (NEACCC)
* Have a pre-incarceration history of substance use disorder
* Have a history of traumatic event exposure and self-report ongoing trauma-related difficulties
* Be within 9 months of release from incarceration
* Expect to reside in Arkansas throughout the study period

Inclusion criteria for prisoners to enroll in the Hybrid Trial in Aim 3 (additional requirements):

* All items listed in "Inclusion criteria for all participants"
* All items listed in "Inclusion criteria for prisoners completing pre-treatment assessments in Aim 3"
* Evidence clinically significant PTSD symptoms during pre-treatment (baseline) assessment per the Structured Clinical Interview for the DSM
* Have a pre-incarceration history of substance use disorder (confirmed by clinical interview)

Exclusion criteria for prisoners to enroll in the Hybrid Trial in Aim 3 (additional requirements):

* Unwilling to consent to randomization
* Unable to provide locator information for post-release assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Post-Incarceration Drug Use | Approximately 3 months after release from incarceration
  Drug use will be examined as both binary responses (abstinence vs. any use) and frequency counts (number of days of use). These variables will be derived from information gained via Timeline Follow-Back Interview.
Change in PTSD Symptoms by Treatment End and 3 Months Post-Release from Incarceration | Pre-treatment assessments will be completed within 4 weeks of treatment start. Post-treatment assessments will be completed within 2 weeks of treatment end. Post-release assessments will be completed approximately 3 months after release from prison.
  PTSD symptoms will be assessed using the 20-item PTSD Checklist (PCL-5). Response options are used to indicate the severity of each PTSD symptom and range from 0 (not at all) to 4 (extremely). Total scores range from 0-80. Lower scores indicate lower levels of PTSD symptoms and therefore a better treatment outcome.

SECONDARY OUTCOMES:
Change in Depression Symptoms by Treatment End and 3 Months Post-Release from Incarceration | Pre-treatment assessments will be completed within 4 weeks of treatment start. Post-treatment assessments will be completed within 2 weeks of treatment end. Post-release assessments will be completed approximately 3 months after release from prison.
  Depression symptoms will be assessed using the Patient Health Questionnaire (PHQ-9). Response options are using to indicate the severity of each symptom of depression and range from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27. Lower scores indicate lower levels of depression symptoms and therefore a better treatment outcome.
Recidivism | 12 months after release from incarceration
  Recidivism will be extracted from administrative incarceration records and examined as both a binary variable (presence or absence of any drug-related recidivism) and frequency counts (number of new drug charges).

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Zielinski, Phd, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - Northeast Arkansas Community Correction Center (NEACCC), Osceola, Arkansas
  - East Central Arkansas Community Correction Center (ECACCC), West Memphis, Arkansas

IPD SHARING:
Plan to Share IPD: Yes
In compliance with NIH's requirement for data sharing, final research data for this project will be made as available as possible upon request while safeguarding the privacy of participants. Individual-level data will be stripped of identifiers and unusual characteristics prior to sharing. A data sharing agreement with the PI will be required.
Supporting Information: Study Protocol, ICF
Time Frame: 12 months after publication of study primary outcome paper.
Access Criteria: Completion of data sharing agreement with PI.

REFERENCES:
- [Derived] Zielinski MJ, Smith MKS, Kaysen D, Selig JP, Zaller ND, Curran G, Kirchner JE. A participant-randomized pilot hybrid II trial of group cognitive processing therapy for incarcerated persons with posttraumatic stress and substance use disorder symptoms: study protocol and rationale. Health Justice. 2022 Oct 1;10(1):30. doi: 10.1186/s40352-022-00192-8. PMID 36181587

DOCUMENTS (1):
  • Informed Consent Form (2022-02-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT04007666/ICF_001.pdf